CLINICAL TRIAL: NCT06312462
Title: A Survey on the Knowledge, Attitudes, and Practices of Students Regarding Schistosomiasis Through a Health Education Model Led by Community Health Volunteers.
Brief Title: Health Education Model Led by Community Health Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pemba Ministry of Health Zanzibar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PembaMoH
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Schistosomiasis; Health Education
Keywords: Schistosomiasis; CHVs; KAP
MeSH Terms: conditions — Schistosomiasis; Health Education

STUDY DESIGN:
Intervention Model Description: This model evaluates the effectiveness of schistosomiasis health education led by community health volunteers by training the volunteers on Pemba Island and having them conduct health education for local students. It also discusses the feasibility of promoting this model in Africa.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHVs Intervention group (Experimental): A group of students who receive schistosomiasis health education intervention led by community health volunteers.
  Interventions: Behavioral: health education
- Control A (No Intervention): A group of students who do not receive schistosomiasis health education intervention led by community health volunteers. The control arm received conventional education.
- Control B (No Intervention): A group of students who do not receive schistosomiasis health education intervention led by community health volunteers. The control arm received conventional education.

INTERVENTIONS:
Behavioral: health education — In the intervention group, we provide schistosomiasis health education to students once a month through community health volunteers for a duration of six months. After that, the community health volunteers no longer visit the school for health education until the completion of a one-year follow-up period.
  Other Names: led by community health volunteers
  Arms: CHVs Intervention group

SUMMARY:
The goal of this intervention study is to investigate the level of knowledge, attitudes, and behaviors of students on schistosomiasis in Pemba Island. It aims to test the effectiveness of establishing a widely applicable Community Health Volunteers model in the Zanzibar region and explore the feasibility of promoting this model in other areas of Africa. This study also aims to provide valuable insights and references for global schistosomiasis prevention and control efforts.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

Conducting a survey to understand the current knowledge levels, attitudes, and relevant health behaviors of Pemba Island students towards schistosomiasis.

Performing qualitative research to analyze the factors influencing students' knowledge, attitudes, and behaviors related to schistosomiasis, as well as observing the facilitators and barriers to conducting health education among student groups, in order to provide a scientific basis for targeted intervention measures.

Testing the effectiveness of establishing a widely applicable community health volunteer model in the Zanzibar region and exploring the feasibility of promoting this model in other regions of Africa, thereby providing insights and references for global schistosomiasis prevention and control efforts.

Participants will select fourth and fifth grade students from two schools located in high-risk schistosomiasis prevalence areas on Pemba Island, with Kilindi Primary School as the intervention group and Shumba Viamboni or Chambani primary school as the control group from Feb 2024 to Feb 2025. Apart from the KAP survey, urine samples will be collected from students three times at least and the prevalence confirmed to compare the effectiveness of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals whose grades fall within the scope of the survey Students who have not received health education intervention on schistosomiasis conducted by community health volunteers Students or parents who agree to sign informed consent and participate in the study Students residing in schistosomiasis-endemic areas

Exclusion Criteria:

* Students whose grades are not within the scope of the survey Students who have already received health education intervention on schistosomiasis Students or parents who refuse to sign informed consent or participate in the study Students who have been diagnosed with other serious illnesses.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 978 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Juma, MSc, Study Chair — NTD office in Pemba
Locations (1):
- Neglected tropical diseases in Pemba, Pemba, CharkChark, Tanzania

RESULTS

PARTICIPANT FLOW:
Groups:
- Control A; Control B: A group of students who do not receive schistosomiasis health education intervention led by community health volunteers, but receive conventional health education.
Period: Overall Study
Arm/Group | CHVs Intervention Group | Control A | Control B
Started | 278 | 324 | 376
Completed | 245 | 295 | 346
Not Completed | 33 | 29 | 30

BASELINE CHARACTERISTICS:
Groups:
- Control A; Control B: A group of students who do not receive schistosomiasis health education intervention led by community health volunteers, but receive conventional health education intervention.
- Total: Total of all reporting groups
Arm/Group | CHVs Intervention Group | Control A | Control B | Total
Number analyzed (Participants) | 245 | 295 | 346 | 886
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.75 (1.441) | 11.98 (1.370) | 11.97 (1.368) | 11.87 (1.405)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 182 | 208 | 535
  Male | 100 | 113 | 138 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 245 | 295 | 346 | 886

OUTCOME MEASURES:

1. Primary Outcome: Change in Infection Rate
Description: For biological sample collection, students provided first-morning urine samples (30-50 mL) in sterile, pre-labeled wide-mouth containers under teacher supervision to ensure protocol adherence. Certified laboratory technicians performed standardized filtration and microscopic analysis to detect S. haematobium eggs. All egg counts were initially recorded manually, then entered into a Microsoft Excel database using dual-entry verification to maintain data integrity. Infection intensity classified by WHO criteria (light: 1-49 eggs/10ml urine; heavy: ≥ 50 eggs/10ml urine)
Time Frame: before the intervention, six months after the intervention, and at the end of the one-year observation period
Measure: Number; unit: Number of Participants with S. haematobi
Groups:
- Control A; Control B: A group of students who do not receive schistosomiasis health education intervention led by community health volunteers.
Arm/Group | CHVs Intervention Group | Control A | Control B
Number analyzed (Participants) | 245 | 295 | 346
Number of Participants with S. haematobi
  baseline(T1) | 47 | 35 | 3
  six months after the intervention（T2） | 6 | 4 | 3
  at the end of the one-year observation period（T3） | 2 | 3 | 5

2. Primary Outcome: Change in Knowledge Scores
Description: Measurement Tool: "Schistosomiasis Knowledge Questionnaire" Description: This questionnaire assesses the knowledge level of students regarding schistosomiasis.
  Scale Title: Schistosomiasis Knowledge Questionnaire Range: Minimum value: 0, Maximum value: 10 Interpretation: Higher scores indicate a better understanding of schistosomiasis
Time Frame: before the intervention, six months after the intervention, and at the end of the one-year observation period
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | CHVs Intervention Group | Control A | Control B
Number analyzed (Participants) | 245 | 295 | 346
Scores
  before the intervention（T1） | 6.11 (1.79) | 6.42 (1.56) | 6.27 (1.47)
  six months after the intervention（T2） | 7.13 (1.44) | 6.62 (1.32) | 7.22 (1.23)
  at the end of the one-year observation period（T3） | 7.11 (1.35) | 6.56 (1.70) | 6.62 (1.56)

3. Primary Outcome: Attitudes Changes
Description: Measurement Tool: "Schistosomiasis Attitudes Questionnaire" Description: This questionnaire assesses the attitudes level of students regarding schistosomiasis.
  Scale Title: Schistosomiasis Attitudes Questionnaire Range: Minimum value: 11, Maximum value: 55 Interpretation: Higher scores indicate more positive attitudes related to schistosomiasis
Time Frame: before the intervention, six months after the intervention, and at the end of the one-year observation period
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | CHVs Intervention Group | Control A | Control B
Number analyzed (Participants) | 245 | 295 | 346
Scores
  before the intervention（T1） | 38.02 (8.49) | 39.06 (8.96) | 39.37 (9.98)
  six months after the intervention（T2） | 41.2 (8.66) | 41.24 (8.15) | 42.55 (8.85)
  at the end of the one-year observation period（T3） | 43.58 (8.95) | 41.39 (8.58) | 41.44 (10.68)

4. Primary Outcome: Behaviors Changes
Description: Measurement Tool: "Schistosomiasis Behaviors Questionnaire" Description: This questionnaire assesses the behaviors level of students regarding schistosomiasis.
  Scale Title: Schistosomiasis Behaviors Questionnaire Range: Minimum value:10 , Maximum value:30 Interpretation: Higher scores indicate more positive behaviors related to schistosomiasis
Time Frame: before the intervention, six months after the intervention, and at the end of the one-year observation period
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | CHVs Intervention Group | Control A | Control B
Number analyzed (Participants) | 245 | 295 | 346
Scores
  before the intervention（T1） | 19.05 (2.74) | 19.35 (2.87) | 19.43 (2.62)
  six months after the intervention（T2） | 20.56 (2.84) | 20.25 (2.64) | 19.77 (2.59)
  at the end of the one-year observation period（T3） | 20.7 (2.912) | 20.14 (2.66) | 19.6 (2.6)

ADVERSE EVENTS:
Time Frame: During the two subsequent follow-up waves : six months after the intervention(2024.08.30): strict individual self-matching and accounting for attrition (school transfers, absenteeism, and incomplete samples; at the end of the one-year observation period(2025.02.27): strict individual self-matching and accounting for attrition (school transfers, absenteeism, and incomplete samples
Description: This research does not involve drug studies and will not endanger the lives of the participants.
Arm/Group | CHVs Intervention Group | Control A | Control B
All-Cause Mortality (participants affected / at risk) | 0/278 | 0/324 | 0/376
Serious Adverse Events (participants affected / at risk) | 0/278 | 0/324 | 0/376
Other Adverse Events (participants affected / at risk) | 33/278 | 29/324 | 30/376
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHVs Intervention Group (N=278) | Control A (N=324) | Control B (N=376)
school transfers (Investigations) | 3 (33) | 2 (29) | 4 (30) — This research does not involve drug studies and will not endanger the lives of the participants. Adverse events were present due to the following circumstances: school transfers, absenteeism, and incomplete samples.
absenteeism (Investigations) | 5 (33) | 4 (29) | 6 (30)
incomplete samples (Investigations) | 25 (33) | 23 (29) | 20 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT06312462/Prot_SAP_000.pdf